Title: Education Time Influence on Exercise-Induced Hypoalgesia

NCT 05658224 Date: 7/10/2023

# CONSENT FORM TO PARTICIPATE IN A RESEARCH STUDY The University of South Dakota

**TITLE:** Grid Localization Testing effects of different grid sizes

**PRINCIPAL INVESTIGATOR:** Dr. Kory Zimney, 605-658-6373, kory.zimney@usd.edu

**Department:** Physical Therapy

## **Invitation to be Part of a Research Study**

You are invited to participate in a research study. You can participate if you are:

- Age 18-64
- A current USD student
- Do <u>NOT</u> have any back pain or sensory deficits

Taking part in this research project is voluntary. Please take time to read this entire form and ask questions before deciding whether to take part in this research project.

## What is this study about and why are we doing it?

We are doing this study to investigate different grid size effects on accuracy with a Grid Localization Test. A Grid Localization Test is a sensory test performed by healthcare professionals to help determine tactile acuity in individuals. Tactile acuity is a measure of the sensitivity of your touch sensory system. About 40 people will take part in this research.

## What will happen if you take part in this study?

If you agree to take part in this study, you will be asked to lie on your stomach and expose the skin on your back. Investigators will touch your back in different spots according to the grid that is placed on your back. You will try and determine where each touch is occurring. You will do this three times with different size grids for each trial. It will take approximately 30 minutes for the entire testing, and you only need to do one session.

### Your Participation in this Study is Voluntary

It is up to you to decide whether to be in this research study. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to answer any questions you do not want to answer. If you decide to withdraw before this study is completed, your data will be destroyed and not used in the study. Your participation will be kept confidential with only the student investigators aware of who is tested. Your data will be deidentified prior to the PI seeing the data. Your participation or lack of participation will not affect your grade or standing in the class or PT program in any way.

#### What risks might result from being in this study?

There are some risks you might experience from being in this study. They are psychological strain or frustration and performance anxiety. To minimize these risks, we will not inform you of your accuracy score during the testing to create any undue performance anxiety of a set score to achieve. The psychological strain of recognizing the touch area or frustration if unable to determine location can occur. You will be reminded by the investigators that it is normal to not be able to always recognize where the touch is occurring. These risks are not viewed as being in excess of your experiences in everyday life.

## What are the potential benefits from this study?

Although you will not directly benefit from being in this study, others might benefit because we will improve our understanding of developing this sensory test further.

## How will we protect your information?

The records of this study will be kept confidential to the extent permitted by law. Any report published with the results of this study will not include any information that could identify you. We will protect the confidentiality of the research data by only recording a non-identifiable code to your research data.

It is possible that our study data will need to be reviewed by people at the University of South Dakota and other agencies as required by law or allowed by federal regulations.

## How will my information be used after the study?

After this study is complete, your deidentified data may be stored indefinitely in secure cloud storage and shared with other researchers through an open access repository without asking for additional consent from you. Your deidentified data will NOT include your name or other personal information that could directly identify you.

#### Contact Information for the Study Team and Questions about the Research

The researchers conducting this study are Dr. Kory Zimney, Jhett Cihak, Taylor Janovy, and Grace Robison. You may ask any questions you have now. If you later have questions, concerns, or complaints about the research please contact Dr. Kory Zimney at 605-658-6373, <a href="mailto:kory.zimney@usd.edu">kory.zimney@usd.edu</a>

If you have problems, complaints, or concerns about the research, questions regarding your rights as a research subject, or if you want to talk with someone independent of the research team, you may contact The University of South Dakota Office of Human Subjects Protection at irb@usd.edu or (605) 658-3743.

#### **Your Consent**

Before agreeing to be part of the research, please be sure that you understand what the study is about. You should keep a copy of this document for your records. If you have any questions about the study later, you can contact the study team using the information provided above.

| I understand that by signing below, I volunteer waiving any legal rights. I have been provided | 1 1 | nd that I am not |
|---|---|---|
| Subject's Name: | | |
| Signature of Subject | Date | |